CLINICAL TRIAL: NCT06688552
Title: Comparison of Acute Effects of Traditional Set and Drop Set Training Methods on Fatigue Levels and Proprioceptive Sensory Mechanism in Bodybuilding Athletes
Brief Title: Comparison of Acute Effects of Traditional and Drop Set Training on Fatigue and Proprioception in Bodybuilding Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giresun University (Other)
Responsible Party: Principal Investigator, Nihat Sarıalioğlu, Asst. Prof., Giresun University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GRU-SBF-NS-02
Record Dates: First submitted 2024-11-11; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Fatigue Intensity; Proprioception
Keywords: drop set; traditional set; fatigue; proprioception
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: This study is a randomised controlled (parallel group) experimental study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional set training (Active Comparator): Traditional set method and drop set method are widely used training methods in bodybuilding. Studies have shown that these methods have similar effects on muscle hypertrophy, increasing lean body mass and other metabolic variables when applied in equal volumes. However, there is no comparative study on the effects of these methods on fatigue and proprioceptive mechanism. In this context, it is thought that it is important to reveal the effects of traditional and drop set training methods on these two variables in order to take necessary measures to protect athlete health and improve athlete performance.
  Interventions: Other: Proprioception Measurements; Other: Fatigue Measurement
- Drop set training (Active Comparator): Traditional set method and drop set method are widely used training methods in bodybuilding. Studies have shown that these methods have similar effects on muscle hypertrophy, increasing lean body mass and other metabolic variables when applied in equal volumes. However, there is no comparative study on the effects of these methods on fatigue and proprioceptive mechanism. In this context, it is thought that it is important to reveal the effects of traditional and drop set training methods on these two variables in order to take necessary measures to protect athlete health and improve athlete performance.
  Interventions: Other: Proprioception Measurements; Other: Fatigue Measurement

INTERVENTIONS:
Other: Proprioception Measurements — Laser cursor-assisted angle repetition test was used for proprioception assessment. A coordinate plane with different movement angles was fixed on a wall and the person was positioned 1 meter from this wall. The laser pointer was fixed on the person's arm for shoulder proprioception measurement, 5 cm above the elbow to avoid being affected by other joints, 5 cm above the person's wrist for elbow joint proprioception and fixed on the person's second metatarsal bone for wrist proprioception.
Other: Fatigue Measurement — Myoton PRO® (Myoton AS, Tallinn, Estonia) muscle palpation device was used to assess fatigue, and the dynamic stiffness parameter was taken as the basis. The stiffness value is calculated as the maximum acceleration (N/m) of oscillation and deformation in the tissue sensed by the transducer (Chen et al., 2017). The increase in muscle dynamic stiffness has been associated with fatigue level (Klich et al., 2019; Shitova et al., 2020; Wang, 2017). Before the measurement, the athletes' pectoralis major, deltoideus and triceps brachii muscle reference points were determined and marked, and measurements were taken over these points. The athletes were asked to keep their muscles relaxed throughout the measurement in order not to affect the tissue stiffness and the application was performed at room temperature.

SUMMARY:
To compare the acute effects of traditional and drop set training methods on fatigue levels and proprioceptive sensory mechanisms in bodybuilding athletes.

DETAILED DESCRIPTION:
A total of 28 male bodybuilding athletes with an average age of 25.53 years from Giresun and Ordu provinces participated in the study voluntarily. The participants were randomly divided into two groups as traditional training group (GS) (n=14) and drop set training group (DS) (n=14). Borg CR10 Scale and myotonometric measurements (Myoton Pro muscle palpation device) were used to assess fatigue. Myotonometric measurements were performed on the pectoralis major, triceps brachii and deltoideus muscles. Proprioception characteristics were evaluated in four parameters: shoulder flexion, shoulder abduction, elbow flexion and wrist flexion using laser cursor-assisted angle repetition test.

After the application, fatigue levels in pectoralis major, triceps brachii, Borg CR10 parameters and proprioception errors in shoulder flexion, elbow flexion, wrist flexion parameters were significantly higher in the traditional set group compared to the drop set group.

ELIGIBILITY:
Inclusion Criteria:

* -Being male.
* Being between the ages of 20-30.
* To have been doing bodybuilding for at least the last five years.

Exclusion Criteria:

* -Having undergone a serious surgical operation within the last year,
* Having used a performance enhancing product that affects the neuromuscular mechanism within the last year,
* In addition, individuals who did not meet the inclusion criteria were excluded from the study.

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Assessment of Demographic and Physical Characteristics | 1 day
  A personal information form was used to obtain demographic information. The height measurements of the participants were made with a wall-mounted holtain stadiometer and body weight measurements were made with a Tanita MC-580 body analyser. BMI was calculated by dividing body weight by the square of height (kg/m2).
Assessment of Proprioception | 1 day
  Laser cursor-assisted angle repetition test was used for proprioception assessment. A coordinate plane with different movement angles was fixed on a wall and the person was positioned 1 meter from this wall. In the next step, the person's eyes were closed to prevent visual control and was asked to repeat the same joint position 3 times. The coordinate point where the individual brought the arm was marked on the coordinate plane and this process was repeated 3 times for shoulder flexion and abduction. The deviations at the given angles were measured on the horizontal (X) and vertical (Y) coordinate axes on the coordinate plane, the amount of linear deviation from the target was calculated using the Pythagorean theorem (√(x^2+y^2 )), and the arithmetic mean of the 3 deviations was recorded.
  Proprioception level= [(√(x^2+y^2 ))+(√(x^2+y^2 ))+(√(x^2+y^2 ))]/3
Assessment of Fatigue | 1 day
  Myoton PRO® (Myoton AS, Tallinn, Estonia) muscle palpation device was used to assess fatigue, and the dynamic stiffness parameter was taken as the basis. The stiffness value is calculated as the maximum acceleration (N/m) of oscillation and deformation in the tissue sensed by the transducer. The increase in muscle dynamic stiffness has been associated with fatigue level. Before the measurement, the athletes' pectoralis major, deltoideus and triceps brachii muscle reference points were determined and marked, and measurements were taken over these points. The athletes were asked to keep their muscles relaxed throughout the measurement in order not to affect the tissue stiffness and the application was performed at room temperature. All measurements were taken with the participants lying on the stretcher and the device was kept upright to minimise the effect of gravity on tissue properties, with three strokes on the reference points of the muscles.

CONTACTS AND LOCATIONS:
Locations (1):
- Giresun University, Giresun, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I don't want my data to be shared.